CLINICAL TRIAL: NCT07285421
Title: Renal and Vascular Phenotypic Characterization of Patients With Enamel Renal Syndrome Due to a Pathogenic Variant of the FAM20A Gene and Pathophysiological Study of Ectopic Calcifications
Acronym: FAM-Cal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation Université de Paris (Unknown); Université de Liège (Other); Institut Necker Enfants Malades (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP240692; 2024-A02589-38 (Other: Agence nationale de sécurité du médicament et des produits de santé); 24.05810.000413 (Other: Commission Nationale des Recherche Impliquant la Personne Humaine)
Record Dates: First submitted 2025-05-28; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Enamel Renal Syndrome
Keywords: FAM20A; enamel renal syndrome
MeSH Terms: conditions — Amelogenesis imperfecta nephrocalcinosis | interventions — Radiography, Panoramic; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteers (Other): The control group will be made up of healthy volunteers, in order to provide a reference population, matched for the analyses carried out as part of the research, i.e. metabolome, proteome and plasma factors of mineralization.
  Interventions: Diagnostic Test: urinary proteome; Diagnostic Test: urinary metabolome; Diagnostic Test: Evaluation of plasma mineralization factors; Diagnostic Test: Renal ultrasound; Radiation: dental panoramic x-ray; Biological: Blood and urine minimal biology
- Enamel Renal Syndrome Patient (Experimental): The population to be studied is a population of adult patients suffering from enamel renal syndrome with FAM20A mutation.
  Interventions: Diagnostic Test: urinary proteome; Diagnostic Test: urinary metabolome; Diagnostic Test: Evaluation of plasma mineralization factors

INTERVENTIONS:
Diagnostic Test: urinary proteome — Volume 2 ml, with protease inhibitor made one time for each arm of the protocol
Diagnostic Test: urinary metabolome — Sample collected once in the protocol for each arm.
Diagnostic Test: Evaluation of plasma mineralization factors — Complementary plasma analysis during another blood sample collection for both arms
  Other Names: Propensity score; Osteoprotegerin; dp-uc MGP; Fetuin A
Diagnostic Test: Renal ultrasound — Verification of normal renal morphology, absence of nephrocalcinosis
  Arms: Healthy volunteers
Radiation: dental panoramic x-ray — Verification of normal dentition
  Arms: Healthy volunteers
Biological: Blood and urine minimal biology — Fasting blood: creatinine, blood ions (Na + K + Cl + CO2 + Proteins), calcium, phosphate, CBC (Complete Blood Count), liver function tests, lipid profile); Morning fasting urine: creatinine, calcium, phosphate, protein, urinalysis (ECBU)
  Arms: Healthy volunteers

SUMMARY:
In the research, the investigators will characterize the renal and vascular damage and look for factors favoring the formation of calcification induced by enamel renal syndrome.

Patients will undergo four investigations, as part of their routine care, to assess their renal impairment. Each investigation will require a day in the Physiology Department of the George Pompidou European Hospital.

The 4 tests are designed to

* precisely measure your renal filtration capacity,
* evaluate your body's calcium and phosphate regulation,
* evaluate your capacity to regulate the elimination of water from the body
* assess your body's ability to regulate "acid" intake. As part of the research, an additional 20 ml blood sample and a urine sample will be taken during the other samples taken as part of routine care.

Healthy volunteers will undergo blood and urine tests, dental X-rays and renal ultrasound. For healthy volunteers, the aim of the dental X-ray and renal ultrasound is to check that there are no dental or renal abnormalities, so as to rule out not only email-rein syndrome, but also any dental or renal abnormalities that might resemble it. The aim of blood and urine sampling is to measure various molecules that promote calcification or inhibit the calcification process, so as to be able to compare results obtained in healthy subjects with those obtained in patients with enamel renal syndrome. Each healthy subject will be selected to be matched by age and sex to each of the patients included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Informed patient who does not object to participating in the study
* Age ≥ 18 years
* Be affiliated to a social security scheme or be a beneficiary of such a scheme
* Able to understand the interest and constraints of the study
* Suffering from enamel-renal syndrome with a proven pathogenic variant of FAM20A

Exclusion Criteria:

* Pregnancy
* Breast-feeding
* Simultaneous participation in a therapeutic trial
* Patient under guardianship or curatorship
* Patient under court protection or family guardianship
* Patient under AME
* Enamel-renal syndrome with pathogenic variation in a gene other than FAM20A

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
Glomerular filtration rate | Up to 18 months
  Glomerular filtration rate measurement by measure of renal 99mTc-DTPA clearance

SECONDARY OUTCOMES:
Comparison of urine proteome between patients and healthy volunteers | Up to 18 months
  Identification of candidate mechanisms to approach the pathophysiology of ectopic calcifications through the study of the urinary proteome
Maximal urine osmolality | Up to 18 months
  Evaluation of water regulation by water deprivation test, urine collection after deprivation.
Level of dp-uc MGP | Up to 18 months
  Identification of candidate mechanisms for approaching the pathophysiology of ectopic calcifications by assaying plasma inhibitors of biomineralization.
Level of Fetuin A | Up to 18 months
  Identification of candidate mechanisms for approaching the pathophysiology of ectopic calcifications by assaying plasma inhibitors of biomineralization.
Level of Osteoprotegerin | Up to 18 months
  Identification of candidate mechanisms for approaching the pathophysiology of ectopic calcifications by assaying plasma inhibitors of biomineralization.
Propensity score | Up to 18 months
  Identification of candidate mechanisms for approaching the pathophysiology of ectopic calcifications by assaying plasma inhibitors of biomineralization.
Ammonium chloride urine flow | Up to 18 months
  Urine collection to evaluate the acid regulation after oral ammonium chloride load test.
calciuria rate | Up to 18 months
  Urine collection in order to evaluate calcium regulation.
Ratio TmPi/DFG | Up to 18 months
  Blood and urine collection in order to evaluate phosphate regulation
Calcium score | Up to 18 months
  Thoracic, abdominal and pelvic scan perform in order to evaluate vascular calcium content.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - HEGP - clinical investigation center, Paris
  - HEGP - physiology department, Paris

IPD SHARING:
Plan to Share IPD: Yes
The deidentified individual participant data (IPD) that support the results reported in publications may be shared. Additionally, the IPD outlined in the protocol for a planned meta-analysis may also be made available. A data dictionary defining each field will be made available concurrently with the data transmission.
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing requires approval from both the sponsor and the Principal Investigator (PI), contingent upon a scientific project and the PI team's scientific contribution. The founder may also participate in the decision-making process.
  Teams seeking to acquire IPD must engage with the sponsor and the IP team to discuss the scientific (and commercial) objectives, the specific IPD required, the preferred data transmission format, and the proposed timeline. The necessity to inform patients about data sharing or the obligation to undertake procedures with data protection authorities will be evaluated.
  The provision of data through the secure institutional tools of the sponsor AP-HP will be prioritized.
  Technical feasibility and financial support considerations will precede the obligatory formalization of a contract, including detailed description of data processing and general and specific security measures.
  The processing must adhere to the European General Data Protection Regulation